CLINICAL TRIAL: NCT06779422
Title: Artificial Intelligence-driven, Chatbot-assisted Acceptance and Commitment Therapy (Pai.ACT) for Parents of Young Children With Neurodevelopmental Disorders: A Randomised Controlled Trial
Brief Title: Pai.ACT - An Artificial Intelligence Driven Chatbot Assisted ACT (Full Scale RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Social Welfare Department, Hong Kong (Other Government); Hong Kong Christian Service (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14600024
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Neurodevelopmental Disorders; Autism Spectrum Disorder (ASD); Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: Parenting Stress; Acceptance and Commitment Therapy; Depression; Anxiety; Psychological flexibility; Psychological Interventions; Smartphone-delivered Therapy; Mental well-being; Hong Kong
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two-arm Randomised Controlled Trial (RCT) with a repeated-measures parallel-group design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Consented articipants will be randomly assigned to either the Pai.ACT Group or Control Group in a 1:1 ratio, using the permuted block size of 6 stratified by child's age (2-3, 4-6) through sequentially numbered, opaque and sealed envelopes with number cards (1=intervention, 2=control). A separate set of random numbers, concealed from the research team and RAs, will be generated by a statistician. Clerical staff uninvolved in the project will administer the randomisation. RA-1, blinded to subject selection, will open the envelopes only after informed consent and baseline assessments are completed. Parents in both study groups will receive a secure e-link for their assigned intervention, accessible via unique login credentials that can tie to their mobile device's ID, as well as a once-weekly reminder to prompt participation. Pai.ACT features content-locking to prevent screen-recording or sharing of audio and video contents to other parents. RA-2, also blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pai.ACT Group (Experimental): Parents allocated to this experimental group will gain complete access to the Pai.ACT mobile app, featuring a 6-week, AI chatbot-assisted Focused ACT intervention for Cantonese-speaking parents of children with NDD, plus one 30-45-minute, individual-based videoconferencing booster session via the Pai.ACT app, mirroring the final session of Focused ACT.
  Interventions: Behavioral: Pai.ACT
- Control Group (Other): Parents in the Control group will receive 6-week mobile-based e-reading modules (30-45 mins of completion/module) about positive parenting advice as recommended by the Child Assessment Services under the Department of Health, plus one 30-45 minute videoconferencing session led by another experienced counsellor for content revision. No access to AI chatbot/ACT modules will be granted.
  Interventions: Other: Positive parenting advice

INTERVENTIONS:
Behavioral: Pai.ACT — The Pai.ACT mobile app is an innovative therapeutic tool that utilizes Acceptance and Commitment Therapy (ACT). It integrates a sophisticated algorithm to analyze self-reported data and conversation texts when the user interacts with the AI chatbot and identifies what psychological inflexibility processes are required to be the most essential to be addressed for process-matched ACT interventions. These interventions, including self-help modules and experiential exercises, are enhanced with dynamic animations and audio metaphors (see NCT06086951). The contents of Pai.ACT is underpinned by: (i) the core principles of Focused ACT, (ii) our validated Focused ACT protocol used in our ongoing Focused ACT trial (see NCT05803252), and (iii) our validated ACT protocols, established since 2019, that address psychological challenges specific to the Chinese parenting context (e.g., affiliate stigma, internalisation of external criticism, self-blame) through a 4-to-6 week of ACT.
  Arms: Pai.ACT Group
Other: Positive parenting advice — Positive parenting advice is recommended by the Child Assessment Services under the Department of Health, and videoconferencing session(s) led by another experienced counsellor for content revision. No access to AI chatbot/ACT modules will be granted.
  Arms: Control Group

SUMMARY:
Interventions for parents of children with NDD face two pivotal challenges. Firstly, many overlook the consequential influence of parenting stress, symptoms of parental anxiety and depression on the well-being of parent-child dyads. Though some address parenting stress, they fall short of considering comprehensive health outcomes. Secondly, current evidence has supported ACT as an empirically validated, transdiagnostic psychotherapeutic intervention for parents with dual benefits for the parent-child dyads, but the treatment delivery (e.g., group-based and guided online approaches) is primarily in-person, demanding the presence of expert personnel in every session, limiting its scalability and accessibility. Unlike other psychotherapies like CBT and mindfulness, conventional ACT sessions often adopt a 'one-size-fits-all' strategy, using standardised and pre-packed exercises lacking the personalisation necessary to address individual variations in psychological inflexibility.

Leveraging our available innovation, Pai.ACT, an AI-driven chatbot adopting the Focused ACT approach, seeks to offer personalised and scalable mental health solutions for Chinese-speaking parents of NDD children. With our encouraging preliminary data supporting our pre-trained NLP model's accuracy and Pai.ACT's feasibility, the investigators propose to examine Pai.ACT in a full-scale clinical trial. The study will examine the following research questions:

1. Is Pai.ACT more effective than positive parenting advice for reducing parenting stress (primary outcome for parents) of parents and the emotional and behavioural symptoms of their young children with NDD (primary outcome for children) over the 12-month post-intervention follow-up?
2. Is Pai.ACT more effective than positive parenting advice for reducing symptoms of depression and anxiety, improving parental psychological flexibility and parenting behaviour over the 12-month post-intervention follow-up?
3. Is Pai.ACT more effective than positive parenting advice for reducing the use of healthcare and rehabilitation services in children with NDD over the 12-month post-intervention follow-up?
4. What are the perceived benefits, satisfaction, strengths, and limitations of Pai.ACT from the parents' perspectives?

DETAILED DESCRIPTION:
Neurodevelopmental disorders (NDD) refer to a diverse group of conditions that commonly emerge during early childhood and are characterized by developmental deficits, resulting in challenges to personal, social, and/or occupational functioning. In Hong Kong, attention-deficit/ hyperactivity disorder (ADHD), autism spectrum disorder (ASD) and developmental delay are the most common types of NDD, and they often co-occur. According to the latest statistical report by the Education Bureau, it is estimated that at least 73,112 pre-schoolers and school-aged children are diagnosed with NDD and are currently receiving special education and/or healthcare services. However, interventions for parents of children with NDD face two pivotal challenges. Firstly, many overlook the consequential influence of parenting stress, symptoms of parental anxiety and depression on the well-being of parent-child dyads. Though some address parenting stress, they fall short of considering comprehensive health outcomes. Secondly, current evidence has supported ACT as an empirically validated, transdiagnostic psychotherapeutic intervention for parents with dual benefits for the parent-child dyads, but the treatment delivery (e.g., group-based and guided online approaches) is primarily in-person, demanding the presence of expert personnel in every session, limiting its scalability and accessibility. Unlike other psychotherapies like CBT and mindfulness, conventional ACT sessions often do not adopt a 'one-size-fits-all' strategy, using standardised and pre-packed exercises lacking the personalisation necessary to address individual variations in psychological inflexibility. Therefore, our team has led multiple ACT trials for parents, both locally and internationally. Leveraging our available innovation, Pai.ACT, an AI-driven chatbot adopting the Focused ACT approach, seeks to offer personalised and scalable mental health solutions for Cantonese-speaking parents of NDD children. With our encouraging preliminary data supporting our pre-trained NLP model's accuracy and Pai.ACT's feasibility, the investigators propose to examine Pai.ACT in a full-scale clinical trial.

Acceptance and Commitment Therapy Acceptance and Commitment Therapy (ACT) has recently emerged as a promising, low-intense psychotherapy for addressing parenting challenges. By practising core ACT skills like cognitive defusion, acceptance, and value clarification, parents can better navigate difficult parenting experiences and reconnect with their caregiving qualities. Extensive research supports the effectiveness of ACT in improving psychological wellbeing and reducing somatic complaints across diverse populations. Recent clinical trials targeting paediatric conditions such as asthma, ASD cerebral palsy, and acquired brain injury have shown significant reductions in parenting stress, depression, and anxiety symptoms. However, in-person delivery of ACT poses barriers, particularly for parents of children with special needs. Utilising smartphones allows convenient access to ACT interventions, accommodating parental caregiving responsibilities, overcoming traditional treatment limitations, and reducing resource requirements for healthcare systems. Studies indicate parents' interest and willingness to incorporate technology into their care, with smartphone-based ACT interventions demonstrating positive effects on parental wellbeing, psychological flexibility, mindfulness skills, and children's quality of life. Yet, challenges persist in maintaining user engagement in these publicly accessible mental health initiatives, with over 70% of individuals discontinuing use shortly after downloading.

Pai.ACT Pai.ACT is a smartphone application that enhances mental health support for parents of children with special healthcare needs in Hong Kong. Integrating Acceptance and Commitment Therapy (ACT) with advanced natural language processing, it offers personalized therapeutic communications in Chinese. Developed through funding from the Innovation and Technology Fund for Better Living (FBL), detailed at https://fbl.itc.gov.hk/approvedproject/1045/ViewPublishItem, Pai.ACT was informed by extensive research including over 19,000 annotated ACT texts. Its patented deep-learning model, trained on a vast collection of Chinese therapeutic dialogues, achieves over 80% accuracy in identifying psychological inflexibility, surpassing existing large language models. This enables Pai.ACT to emulate the assessment skills and empathetic responses of trained ACT practitioners, providing users with tailored and scalable mental health assessments and interventions. Pai.ACT also utilises a sophisticated voice-to-text chatbot system that mimics interactions with ACT-trained counsellors, providing personalised self-guided mental health assessments and interventions.

STUDY AIMS

1. To examine the effectiveness of an AI-driven chatbot, smartphone-enabled Acceptance and Commitment Therapy (ACT) approach, referred to as Pai.ACT, compared to positive parenting advice in reducing parenting stress (primary outcome for parents) of parents and the emotional and behavioural symptoms of their young children with NDD (primary outcome for children) over the 12-month post-intervention follow-up.
2. To assess the effectiveness of Pai.ACT compared to positive parenting advice in reducing symptoms of depression and anxiety, improving parental psychological flexibility and parenting behaviour over the 12-month post-intervention follow-up.
3. To examine the effectiveness of Pai.ACT compared to positive parenting advice in reducing the use of healthcare and rehabilitation services in children with neurodevelopmental disorders over the 12-month post-intervention follow-up.
4. To explore the perceived benefits, satisfaction, strengths, and limitations of Pai.ACT from the parents' perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers who are Cantonese-speaking Hong Kong residents.
* Parents aged ≥21 years.
* Primary caregivers who adopt the responsibility of taking care of the child.
* Living together with the child and having smartphone devices for daily access to the internet.
* Parent's children should be with following criteria:

  i) Aged 2-6 years. ii) Received a primary and clinical diagnosis/suspected diagnosis of NDD as indicated in the clinical records according to the DSM-5 criteria. (e.g., ASD, ADHD, developmental delay) iii) Registered for Social Welfare Department subvented Onsite Pre-school Rehabilitation Services.

Exclusion Criteria:

* Parents diagnosed with severe mental illnesses.
* Parents with learning, cognitive, language, communication impairments or other debilitating conditions. (e.g., hearing or vision impairment) that could impede full participation in the study)
* Parents currently participating in /under the evaluation of other psychosocial, psychoeducation or parenting programmes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-02-13 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Parenting stress will be evaluated utilising the Parenting Stress Index-Short Form (PSI-SF), comprising 36 items on a 5-point Likert scale. The PSI-SF assesses stress across three dimensions: parental distress, dysfunctional parent-child interaction, and challenging child behaviour, with a higher total score reflecting greater stress. The Chinese version of the PSI-SF has demonstrated robust convergent and discriminant validity, as well as internal consistency (α = .79-.88) in a Chinese parental cohort.
Child Emotional and Behavioural Symptoms | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Child emotional and behavioural symptoms will be evaluated using the Strengths and Difficulties Questionnaire (SDQ), which consists of 25 items on a 3-point Likert scale. The SDQ, a parent-reported measure, assesses five domains: emotional symptoms, conduct issues, hyperactivity/inattention, peer-related problems, and prosocial behaviour, with a higher total score reflecting more symptoms. The Chinese version of the SDQ has shown satisfactory test-retest reliability (ICC = .75-.86) and discriminant validity among Hong Kong parents.

SECONDARY OUTCOMES:
Symptoms of Depression and Anxiety | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Symptoms of parental anxiety and depression will be assessed through the Generalised Anxiety Disorder-7 (GAD-7; 7-item, 4-point Likert scale) and the Patient Health Questionnaire-9 (PHQ-9; 9-item, 4-point Likert Scale), respectively, with high scores reflecting more severe symptoms. Both instruments have demonstrated adequate concurrent validities with other mental health measures (e.g., SF-12) and internal consistencies (α = 0.92 in GAD-7; 0.82 in PHQ-9) in HK samples.
Parental Psychological Flexibility | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Parental psychological flexibility will be measured using the Psyflex questionnaire, a 6-item scale with a 5-point Likert scale. This instrument evaluates six dimensions of psychological flexibility: defusion, acceptance, present-moment contact, self-as-context, values, and committed action, The Psyflex has demonstrated excellent convergent and divergent validity, as well as reliability (Raykov's r = .91). Its Chinese version has been validated in the PI's work.
Parenting Behaviour | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Parenting behaviour will be assessed using the Interpersonal Mindfulness in Parenting Scale (IM-P), a 23-item scale with a 5-point Likert scale. The IM-P assesses adaptive parenting behaviour across four dimensions: present-centred attention, emotional awareness, non-reactivity, and non-judgmental acceptance. The Chinese version of the IM-P has shown adequate convergent validity and internal consistency (α = .70-.84) among Hong Kong parents.
The use of health care and rehabilitation services | Change from baseline to immediate, 3-month, 6-month and 12-month post-intervention
  Utilisation of child healthcare and rehabilitation services, including the types and frequencies of services accessed from both private and public sectors over the preceding 12 months, will be assessed by parental reports and then crosschecked with the records provided by the Onsite Pre-school Rehabilitation Services teams.

IPD SHARING:
Plan to Share IPD: Undecided